CLINICAL TRIAL: NCT07008222
Title: Pain Related to Local Anesthetic Administration for Nexplanon Placement: A Randomized Control Trial of Buffered Lidocaine
Brief Title: Pain Related to Local Anesthetic Administration for Nexplanon Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, MD, MPH, Obstetrics, Gynecology and Reproductive Sciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 812038
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Pain Related to Local Anesthetic Administration for Nexplanon Placement
MeSH Terms: interventions — Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Intervention Model Description: The participant and clinician will be blinded to their randomization. The group assignment will be in a sealed envelope opened by the clinic nurse and administered by the clinician. The envelopes will previously have been filled with group assignments (buffered vs nonbuffered lidocaine groups) and will then be shuffled prior to in-clinic use to determine participant group assignment.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buffered Lidocaine Anesthetic Group (Experimental): will prepare 3cc of buffered lidocaine consisting of 2.7cc of 1% lidocaine and 0.3cc of 8.4% sodium bicarbonate
  Interventions: Combination Product: we will prepare 3cc of buffered lidocaine consisting of 2.7cc of 1% lidocaine and 0.3cc of 8.4% sodium bicarbonate
- Un-buffered Lidocaine Anesthetic Group (Active Comparator): 3cc of unbuffered 1% lidocaine
  Interventions: Other: Unbuffered lidocaine

INTERVENTIONS:
Combination Product: we will prepare 3cc of buffered lidocaine consisting of 2.7cc of 1% lidocaine and 0.3cc of 8.4% sodium bicarbonate — Either 3cc of unbuffered lidocaine (control) or 3cc of buffered 1% lidocaine (intervention) will be prepared and administered by the clinician. In a study investigating buffered lidocaine versus unbuffered lidocaine in intrauterine device insertion, investigators prepared 20cc of buffered lidocaine utilizing 18cc of 1% lidocaine (90%) and 2cc of 8.4% sodium bicarbonate (10%). 3 Thus, we will prepare 3cc of buffered lidocaine consisting of 2.7cc of 1% lidocaine and 0.3cc of 8.4% sodium bicarbonate.
  Arms: Buffered Lidocaine Anesthetic Group
Other: Unbuffered lidocaine — For the control, 3cc of unbuffered lidocaine will be prepared and administered by the clinician.
  Arms: Un-buffered Lidocaine Anesthetic Group

SUMMARY:
This research study is being conducted to see if using buffered lidocaine for Nexplanon placement decreases pain associated with administering local anesthesia compared to unbuffered lidocaine, which is currently used in clinic. Lidocaine is used to stop pain in the nerve fibers in order to decrease pain at the time of the procedure. We want to find out if using buffered lidocaine will decrease discomfort at the time of receiving local anesthesia for Nexplanon insertion.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Women, aged 18-50 who are English or Spanish speaking who present for Nexplanon placement for contraception
* Participants must not have a past medical history of substance use disorders, pain disorders, use of pain medications or are found to be pregnant

Exclusion Criteria:

* Current use of pain medication prior to procedure
* Diagnosed chronic pain condition
* Pregnancy
* Known allergic reactions to components of the local anesthetic
* History of Nexplanon placement
* Current substance use or history of substance use
* Known contraindications to Nexplanon, such as history of breast cancer, Systemic lupus erythematosus with positive (or unknown) antiphospholipid antibodies, unexplained vaginal bleeding, and liver conditions, including hepatocellular adenoma, malignant liver tumor, and decompensated cirrhosis.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Magnitude of pain at time of local anesthesia for Nexplanon placement | Will assess pain immediately upon completion of the respective step (i.e. at completion of administration of local anesthetic)
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) recorded at the time of local anesthetic administration for Nexplanon placement

SECONDARY OUTCOMES:
Anticipated pain, prior to anesthetic administration | Will assess anticipated pain immediately prior to anesthetic administration
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) to describe pain anticipated during procedure prior to anesthetic administration.
Baseline pain | At one point in time occurring at some point from the time of enrollment but prior to Nexplanon placement procedure
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) to describe pain at baseline
Pain with Nexplanon placement | Will assess pain associated with Nexplanon placement immediately upon completion of this step
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) to describe pain experienced specifically with placement of the Nexplanon
Pain associated with overall procedure | Will assess pain associated with overall procedure immediately following conclusion of Nexplanon placement procedure
  Distance (mm) from the left of the 100-mm VAS scale (reflecting magnitude of pain) to describe pain associated with the overall Nexplanon placement procedure.
Patient satisfaction | Following completion of Nexplanon placement procedure but prior to conclusion of the procedural visit.
  Will assess participant satisfaction with pain control associated with Nexplanon placement using a Likert scale. We will utilize questions such as "How did the pain with Nexplanon placement compare to the expected pain?", "Would you choose the same pain control method for future implant insertion? and assessing if participant would recommend to a friend (Would you recommend this pain control method to a friend for Nexplanon placement?).
Overall Nexplanon placement experience | Upon completion of Nexplanon placement procedure but prior to conclusion of procedural visit.
  We will assess patient satisfaction with the overall Nexplanon placement experience utilizing VAS scale (anchors 0 mm = not, 100 mm = extremely satisfied).
Need for additional pain medication | Upon completion of Nexplanon placement procedure but prior to conclusion of procedural visit.
  We will assess need for additional pain medication by assessing whether participants require/request additional pain medication (e.g. Tylenol or ibuprofen) prior to completion of their procedural visit.
Participants belief | Upon completion of Nexplanon placement but prior to conclusion of the procedural visit.
  We will assess participants belief regarding if they were in the intervention or control group (i.e. whether they received buffered versus unbuffered lidocaine for local anesthetic prior to Nexplanon placement).

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD, MPH, Principal Investigator — Obstetrics, Gynecology and Reproduc.ve Sciences, UCSD

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bentsianov SD, Brandi K, Chen P, Shimoni N. A Pilot Study to Understand the Adolescent Pain Experience During Contraceptive Implant Insertion. J Pediatr Adolesc Gynecol. 2021 Aug;34(4):522-524. doi: 10.1016/j.jpag.2021.01.013. Epub 2021 Jan 27. PMID 33515699
- [Background] Nelson AL. Neutralizing pH of lidocaine reduces pain during Norplant system insertion procedure. Contraception. 1995 May;51(5):299-301. doi: 10.1016/0010-7824(95)00078-o. PMID 7628204
- [Background] Mody SK, Farala JP, Jimenez B, Nishikawa M, Ngo LL. Paracervical Block for Intrauterine Device Placement Among Nulliparous Women: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):575-582. doi: 10.1097/AOG.0000000000002790. PMID 30095776
- [Background] Azizkhani R, Forghani M, Maghami-Mehr A, Masomi B. The effects of injections of warmed bicarbonate-buffered Lidocaine as a painkiller for patients with trauma. J Inj Violence Res. 2015 Jul;7(2):87-8. doi: 10.5249/jivr.v7i2.523. Epub 2013 Dec 12. No abstract available. PMID 24879075